CLINICAL TRIAL: NCT05534464
Title: Difference in Digestibility of Three Protein Sources Between Older and Younger Adults as Measured With the Dual Tracer Method
Brief Title: Protein Digestibility in Older and Younger Adults
Acronym: DiGest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Marco Mensink, dr. MR (Marco) Mensink, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL80529.091.22
Record Dates: First submitted 2022-07-05; First posted 2022-09-09 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Ageing
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: Participants will have three test days, each separated by two weeks. The participants will randomly consume one of the three protein sources on each test day respectively.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skimmed milk powder (Experimental): One rumen-fistulated Holstein-Friesian dairy cow in high lactation status will be given 0.6 L deuteriated water 3 times per day for 3 days long. Milk collection will take place twice a day on the fourth and fifth day. Milk will be processed into skimmed milk powder.
  Interventions: Other: Milk
- Sorghum whole grain (Experimental): Sorghum plants are grown in the greenhouse. Those receive deuteriated water for five days with one day in between. On the first day the water has a 25% dilution and the other four days the water has a 5% dilution.
  Interventions: Other: Sorghum
- Black beans (Experimental): Black bean plants are grown in the greenhouse. Those receive deuteriated water for five days with one day in between. On the first day the water has a 25% dilution and the other four days the water has a 5% dilution.
  Interventions: Other: Black beans

INTERVENTIONS:
Other: Milk — Twenty grams of the deuterium (2H) - labelled skimmed milk powder mixed with water will be consumed on one of the three different test days. The meal will be divided in 10 portions, consumed every hour. The 2H-labelled protein source is mixed with free 13C-labelled amino acids as reference. Protein free cookies are served alongside to equal macronutrient composition with the other two protein sources.
  Arms: Skimmed milk powder
Other: Sorghum — Twenty grams of the deuterium (2H) - labelled whole grain sorghum cooked with water will be consumed on one of the three different test days. The meal will be divided in 10 portions, consumed every hour. The 2H-labelled protein source is mixed with free 13C-labelled amino acids as reference.
  Arms: Sorghum whole grain
Other: Black beans — Twenty grams of the deuterium (2H) - labelled black beans cooked with water and mashed into a puree, will be consumed on one of the three different test days. The meal will be divided in 10 portions, consumed every hour. The 2H-labelled protein source is mixed with free 13C-labelled amino acids as reference. A carbohydrate drink is served alongside to equal macronutrient composition with the other two protein sources.
  Arms: Black beans

SUMMARY:
The main goal of this study is to determine the difference in amino acid digestibility of milk, sorghum and black beans between older (65-80 years) and younger (20-35 years) adults using the dual tracer method.

DETAILED DESCRIPTION:
Older adults should meet their amino acid requirements to prevent development of sarcopenia. Dietary protein quality is of importance, as determined by amino acid composition and digestibility of the consumed protein. There is a need to investigate the impact of ageing on amino acid digestibility and thus quality in vivo. The dual tracer method is an indirect, minimal-invasive method to determine amino acid digestibility in humans. It is expected that amino acid digestibility decreases with age and that the effect between age groups is greater for poorly digestible protein sources. In this randomized, cross-over study, the researchers will determine the difference in amino acid digestibility of milk, sorghum and black beans between older (65-80 years) and younger (20-35 years) adults using the dual tracer method. Secondary objectives concern the difference in amino acid kinetics between older and younger adults and the association between gut health plasma markers and amino acid digestibility.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-35 years or 65-80 years
* Body Mass Index (BMI): 20.0 - 30.0 kg/m2
* Veins suitable for blood sampling
* Healthy as assessed with a questionnaire
* Regular and normal Dutch eating habits as assessed with a questionnaire
* Having given written informed consent
* Willing to comply with study procedures
* Accept use of all encoded data, including publication, and the confidential use and storage of all data for 15 years.

Exclusion Criteria:

* Chronic disease, for example:

  * Diabetes mellitus, being treated for high blood glucose or increased fasting blood glucose (> 6.7 mmol/l in finger prick blood)
  * Active cardiovascular disease
  * Hepatic disease (e.g. hepatitis)
  * Renal disease
  * Cancer
  * Bowel disease (e.g. inflammatory bowel disease, ulcers, bleeding)
  * Pancreatitis
* History of medical or surgical events that may affect GI function and the study outcomes, for example:

  * Bariatric surgery
  * Gastrointestinal tract surgery
  * Digestive tract disorder
  * Chewing problems
* Medicine use that interferes with GI function and the study outcomes, for example:

  * Glucose lowering drugs
  * Proton pump inhibitors
  * Laxatives
* Habits that interfere with the study outcomes:

  * Probiotics and/or protein supplement use
  * Smoking
  * Drug abuse
  * Alcohol consumption for men >21 units/week and >4/day and for women >14 units/week and >3/day
  * Following a weight-loss diet, medically prescribed diet or other diet with a low calorie intake or an unbalanced nutrient intake like a vegan or very low carbohydrate diet
  * Moderate to high intense physical activity for more than 5 hours a week
  * Difficulties with eating breakfast in the morning
* Other:

  * Self-reported allergy or intolerance to the tested products (milk, sorghum, black beans)
  * Weight loss of more than 3 kg in the month prior to study screening
  * Being pregnant
  * For men: Hb <8,5 mmol/l and for women: Hb <7,5 mmol/l
  * Recent blood donation (<2 months prior to start of the study)
  * Current participation in other research and <2 months previous participation in other research
  * Not having a general practitioner
  * Not willing to accept information-transfer concerning participation in the study, or information regarding his or her health, like laboratory results and eventual adverse events to and from his general practitioner
  * Working at the department of Human Nutrition and Health at Wageningen University & Research

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Amino acid digestibility of three different protein sources | 1 measurement repeated on 3 test days for 3 protein sources respectively, separated by 2 weeks wash-out
  Ratio between meal and plasma isotope enrichment in amino acids

SECONDARY OUTCOMES:
Linear increase in plasma amino acids of three different protein sources | 11 blood samples during 8 hours, repeated on 3 test days for 3 protein sources respectively, separated by 2 weeks wash-out
  Amino acids in plasma are determined over time. First measure of kinetics is the linear increase or the slope of the curve.
Area under the curve for plasma amino acid concentration of three different protein sources | 11 blood samples during 8 hours, repeated on 3 test days for 3 protein sources respectively, separated by 2 weeks wash-out
  Amino acids in plasma are determined over time. Second measure of kinetics is the area under the curve.
Steady state plasma amino acid concentration of three different protein sources | 11 blood samples during 8 hours, repeated on 3 test days for 3 protein sources respectively, separated by 2 weeks wash-out
  Amino acids in plasma are determined over time. Third measure of kinetics is the steady state concentration or the plateau of the curve.
Plasma gut health markers of the participants in relation to age and amino acid digestibility | 1 blood sample before consumption of the protein source, repeated on 3 test days for 3 protein sources respectively, separated by 2 weeks wash-out
  Four gut health markers in plasma will be measured: kynurenine/tryptophan ratio, citrulline, ornithine, I-FABP.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands